CLINICAL TRIAL: NCT01876108
Title: The Effect of Helicobacter Pylori Eradication on Liver Fat Content in Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: The Effect of Helicobacter Pylori Eradication on Liver Fat Content in Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Raika Jamali, MD, Assistant Professor of Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1392/3/11- 589
Record Dates: First submitted 2013-06-08; First posted 2013-06-12 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Fatty Liver; Liver Dysfunction; Insulin Resistance
Keywords: Steatohepatitis; Helicobacter pylori; Alanine aminotransferase; Aspartate aminotransferase; Fatty Liver; Liver Diseases; Digestive System Diseases
MeSH Terms: conditions — Fatty Liver; Liver Diseases; Insulin Resistance; Digestive System Diseases | interventions — Omeprazole; Amoxicillin; bismuth tripotassium dicitrate; Azithromycin

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H.pylori eradication (Experimental): H.pylori eradication by quadruple antibiotic therapy for two weeks plus obtaining ideal body weight by calorie restriction diet and programmed physical activity.
  Interventions: Drug: H.pylori eradication (Omeprazole, Amoxicillin, Bismuth subcitrate, Azithromycin)
- Lifestyle modification (No Intervention): Obtaining ideal body weight by calorie restriction diet and programmed physical activity

INTERVENTIONS:
Drug: H.pylori eradication (Omeprazole, Amoxicillin, Bismuth subcitrate, Azithromycin) — The regimen consists of Omeprazole (20 mg/BD)+ Amoxicillin (1 g/day)+ Bismuth subcitrate (240 mg/BD)+ Azithromycin (500 mg/BD)for two weeks.
  Other Names: H.pylori treatment
  Arms: H.pylori eradication

SUMMARY:
The role of Helicobacter pylori(HP)in the pathogenesis of non-alcoholic fatty liver disease (NAFLD) is controversial.

DETAILED DESCRIPTION:
This randomized double blind clinical trial was performed in dyspeptic patients with positive antibody to HP and the evidence of fatty liver in ultrasonography. After excluding other causes, participants with persistent elevated serum aminotransferase levels were presumed to have NAFLD. Those with NAFLD liver fat score greater than (-0.64) and positive urea breath test (UBT) were enrolled. They were randomly assigned to lifestyle modification alone or lifestyle modification plus HP eradication groups. Quadruple therapy (omeprazole, amoxicillin, bismuth subcitrate, and clarithromycin) for HP eradication was performed in two weeks. HP eradication was documented by UBT. Liver fat content, fasting serum glucose, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, triglyceride, cholesterol, high and low-density lipoprotein,homeostasis model assessment-insulin resistance(HOMA-IR), and anthropometric measurements (body mass index and waist circumference) were checked at baseline and six months later.

ELIGIBILITY:
Inclusion Criteria:

* dyspeptic patients with positive antibody to H.pylori and
* persistent elevated aminotransferase levels with the evidence of fatty liver in ultrasonography, who were referred to a gastroenterology clinic.

Exclusion Criteria:

* alcohol use (more than 20 gram per day in men and 10 gram per day in women per day),
* heart disease (ischemic or congestive),
* hepatic disease (viral hepatitis, autoimmune hepatitis, wilson disease, hemochromatosis, liver mass lesion),
* renal disease (serum creatinine concentration of > 1.5 mg/dl),
* any severe systemic co-morbidities, neoplasm,
* using any hepatotoxic medication during the past 3 months,
* previous history of peptic ulcer,
* previous history of H.pylori eradication,
* existence of alarm signs (weight loss, dysphagia, anemia, vomiting, positive family history of gastrointestinal cancers), and
* pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline liver fat content at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline liver function tests at 6 months | 6 months

OTHER OUTCOMES:
Change from baseline insulin resistance at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Gastroenterology clinic, Sina Hospital, Tehran, Tehran Province, Iran